CLINICAL TRIAL: NCT02828267
Title: Developing a Brief Negotiational Intervention for Alcohol Use Among Injury Patients in Tanzania
Brief Title: Evaluating a Brief Negotiational Intervention for Alcohol Use Among Injury Patients in Tanzania
Acronym: BNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00062061; K01TW010000 (NIH)
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Use
Keywords: Tanzania; Alcohol Use; Brief Intervention
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This is an feasiblity trial of a three stage adaptive clinical trial. Stage one has three arms (UC, BNI, BNI+ Standard booster). Stage two drops usual care arm. Stage three continues the strongest arm for phase two (which was choosen as BNI + Standard Booster for this feasiblity trial not powered to determine efficacy) and a new arm BNI + Personalized Booster.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors are not privy as to which arm patients were randomized to. Participants obviously are aware if they participate in a discussion and receive texts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): In the Usual Care arm, patients will have standard discharge information and instructions without any further health or wellness instruction
- BNI (Experimental): In the BNI arm, patients will receive a 5-30 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions.
  Interventions: Behavioral: Brief Negotiational Intervention
- BNI plus standard booster (Active Comparator): In the BNI plus standard booster arm, patients will receive the 5-30 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions. Then after discharge patients will receive a test focused on reducing alcohol use to a SMS capable cell phone weekly for a total of 6 months of follow up. The messages will be standard messages for all those in this arm.
  Interventions: Behavioral: Brief Negotiational Intervention; Behavioral: Standard Booster
- BNI plus personalized booster (Active Comparator): In the BNI plus personalized booster arm, patients will receive a 5-30 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions. Then after discharge patients will receive a text focused on reducing alcohol use to a SMS capable cell phone weekly for a total of 6 months of follow up. In the personalized arm, the text sent will be personalized based on information obtained about the patient's reasons for reducing their drinking found in the BNI.
  Interventions: Behavioral: Brief Negotiational Intervention; Behavioral: Personalized Booster

INTERVENTIONS:
Behavioral: Brief Negotiational Intervention — This is a 5-10 minute conversation using the principles of motivational interviewing between the healthcare practioner and the patient to motivate the patient to identify at risk alcohol use and through self-empowerment create a plan to decrease alcohol use.
  Arms: BNI; BNI plus personalized booster; BNI plus standard booster
Behavioral: Standard Booster — This SMS based intervention will be a text to the participant once weekly including motivational statements to try to have patients reduce their alcohol use.
  Arms: BNI plus standard booster
Behavioral: Personalized Booster — This SMS based intervention will be a text to the participant once weekly including motivational statements to try to have patients reduce their alcohol use. Information in this text will be personalized based on the participants specific reasons for reducing their alcohol use rather than a standard text content.
  Arms: BNI plus personalized booster

SUMMARY:
A brief negotiational interview (BNI), administered in an Emergency Department setting for both hazardous and harmful drinkers has been shown to cost-effectively reduce a patient's alcohol intake and re-injury rate up to 3 years post intervention. A BNI is a short (5-30 minute) counseling session administered by non-addiction specialists based on the concepts of the FRAMES model of motivational interviewing. Text based boosters have been proposed to prolong the impact of this intervention, either with a standardized or personalized content. The investigators will conduct a pilot study to test the feasibility of the study protocols, acceptance of the intervention, and patient enrollment and retention rates, as we prepare for a fully powered pragmatic randomized adaptive controlled trial of the intervention for patients seen at the Kilimanjaro Christian Medical Center (KCMC) Emergency Department.(ED)

DETAILED DESCRIPTION:
Research Design: This will be a pilot randomized adaptive feasibility and acceptability trial.

This will be a three stage trial where usual care, brief intervention and brief intervention with standard booster will be in the first stage. The second stage will drop the usual care arm. The third stage will keep an arm in stage two and a new arm, brief intervention with personalized booster. Since this is a feasibility trial, we will advance through potential adaptations, changing the enrollment procedures but not based on effectiveness testing as we are not powered for that endpoint. We have chosen brief intervention with standardized booster to continue in stage 3 to obtain more patient experience with the booster portion of the intervention.

Participants and Recruitment: The investigators will prospectively enroll (n=75, 10 usual care, 20 BNI, 24 BNI + standard booster and 16 BNI + Personalized Booster) patients who present to the KCMC ED for care of acute injuries and meet inclusion and exclusion criteria. Trained research nurses will describe the intervention as a health assessment, and eligible interested participants will be enrolled, provide informed consent and a randomization packet chosen. The research nurses will then administer patient demographic, injury, alcohol use surveys and the intervention if appropriate all lasting less than 45 minutes.

Follow-up Procedures: All groups will provide two phone numbers where participants can be reached in order to facilitate follow-up. All participants will be contacted at 6 weeks, 3 months and 6 months for follow-up survey administration. Follow up surveys are expected to be less than 20 minutes. All patients will be contacted by text message at the conclusion of the study to inform them about availability of the results of the study.

Feasibility Trial Outcomes: Using the RE-AIM framework, we will define the reach (enrollment/ retention), the preliminary effectiveness (reduction in DrInC score), adoption including patient acceptance, implementation (intervention fidelity) and maintance (sustainability features). The investigators will conduct a feasibility assessment subjectively through self-assessments as well as objectively through Event Analyses, understanding causes of deviations from protocol, intervention evaluations and questionnaires.

Study Procedures: To evaluate the study procedures, the investigators will evaluate any protocol deviation events, and compare length of survey times. The investigators will also perform assessments of intervention fidelity through reviewing recorded observations of BNI administration using the BNI Assessment Scale.

Reach: Enrollment and Retention The primary outcome measure will be recruitment and retention rates, anticipated at 30% and 60%, respectively. Secondarily, the investigators will qualitatively assess the inclusion and exclusion criteria, reasons for non-enrollment or non-retention, to the extent possible. Finally, the investigators will administer follow-up questions about compensation procedures in order to improve enrollment or retention.

Effectiveness: We will evaluate the DrInC (Drinker Inventory of Consequences), AUDIT (Alcohol Use Disorder Identification Test) scores, number of drinking days and number of binge drinking days. We are not powered to determine effectiveness, so this is a preliminary effectiveness only.

Adoption: We will evaluate patient acceptance and perception of effectiveness for the adoption of this intervention. The investigators will assess acceptability of participation in the trial and intervention through questions administered after the final follow-up time point for both the research team as well as participants. This will include assessment about the length of surveys, and method and quantity of follow-up.

Implementation: We will evaluate implementation preparedness with an evaluation of the time burden of the BNI, and intervention fidelity both for the BNI, and SMS boosters but also trial protocols.

Maintenance: We will determine sustainability through the burden of administration of the BNI as perceived by research nurses administering the intervention, the attitudes towards effectiveness of interventionists and participants, the cost and feasibility of this type of this adaptive clinical trial in this setting.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* be clinically sober at the time of enrollment
* have capacity to give informed consent
* converse in the local language Swahili or in English
* have either:

  * reported ingesting alcohol in the 6 hours prior to injury,
  * have a positive breathalyzer test, or
  * have an Alcohol Use Disorder Identification Test with a score of ≥8.

Exclusion Criteria:

* <18 years of age
* being clinically intoxicated
* being injured so severely that participants do not have the capacity to give informed consent
* not able to converse in Swahili or English

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Staton, MD, MSc, Principal Investigator — Duke University
Locations (1):
- Kilimanjaro Christian Medical Center, Moshi, Tanzania

REFERENCES:
- [Derived] Staton CA, Agnihotri D, Phillips AJ, Ngowi K, Huo L, Boshe J, Sakita F, Tupetz A, Suffoletto B, Mmbaga BT, Vissoci JRN. Development of culturally-appropriate text message booster content to follow a brief intervention focused on reducing alcohol related harms for injury patients in Moshi, Tanzania. PLOS Glob Public Health. 2024 Jul 25;4(7):e0002717. doi: 10.1371/journal.pgph.0002717. eCollection 2024. PMID 39052647
- [Derived] Staton CA, Friedman K, Phillips AJ, Minnig MC, Sakita FM, Ngowi KM, Suffoletto B, Hirshon JM, Swahn M, Mmbaga BT, Vissoci JRN. Feasibility of a pragmatic randomized adaptive clinical trial to evaluate a brief negotiational interview for harmful and hazardous alcohol use in Moshi, Tanzania. PLoS One. 2023 Aug 3;18(8):e0288458. doi: 10.1371/journal.pone.0288458. eCollection 2023. PMID 37535693

RESULTS

PARTICIPANT FLOW:
Groups:
- Brief Negotiational Interview (BNI): In the BNI arm, patients will receive a 5-10 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions.
  Brief Negotiational Intervention: This is a 5-10 minute conversation using the principles of motivational interviewing between the healthcare practioner and the patient to motivate the patient to identify at risk alcohol use and through self-empowerment create a plan to decrease alcohol use.
- BNI Plus Standard Booster: In the BNI plus standard booster arm, patients will receive a 5-10 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions. Then after discharge patients will receive a test focused on reducing alcohol use to a SMS capable cell phone weekly for a total of 6 months of follow up. The messages will be standard messages for all those in this arm.
  Brief Negotiational Intervention: This is a 5-10 minute conversation using the principles of motivational interviewing between the healthcare practioner and the patient to motivate the patient to identify at risk alcohol use and through self-empowerment create a plan to decrease alcohol use.
  Standard Booster: This SMS based intervention will be a text to the participant once weekly including motivational statements to try to have patients reduce their alcohol use.
- BNI Plus Personalized Booster: In the BNI plus personalized booster arm, patients will receive a 5-10 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions. Then after discharge patients will receive a test focused on reducing alcohol use to a SMS capable cell phone weekly for a total of 6 months of follow up. In the personalized arm, the text sent will be personalized based on information obtained about the patient's reasons for reducing their drinking found in the BNI.
  Brief Negotiational Intervention: This is a 5-10 minute conversation using the principles of motivational interviewing between the healthcare practioner and the patient to motivate the patient to identify at risk alcohol use and through self-empowerment create a plan to decrease alcohol use.
  Personalized Booster: This SMS based intervention will be a text to the participant once weekly including motivational statements to try to have patients reduce their alcohol use. Information in this text will be personalized based on the participants specific reasons for reducing their alcohol use rather than a standard text content.
Period: Overall Study
Arm/Group | Usual Care | Brief Negotiational Interview (BNI) | BNI Plus Standard Booster | BNI Plus Personalized Booster
Started | 10 | 21 | 24 | 20
Completed | 10 | 21 | 24 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Brief Negotiational Interview (BNI) | BNI Plus Standard Booster | BNI Plus Personalized Booster | Total
Number analyzed (Participants) | 10 | 21 | 24 | 20 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (12.8) | 40.6 (13.8) | 36.6 (14.5) | 31.4 (11.8) | 36.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 10 | 19 | 23 | 20 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 21 | 24 | 20 | 75
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 10 | 21 | 24 | 20 | 75
Drinker Inventory of Consequences (DrInC) [Mean (Standard Deviation); unit: score on a scale] — The DrInC is a self-administered 50-item questionnaire designed to measure adverse consequences of alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. Scales are combined to assess total adverse consequences, with higher scores indicating more adverse consequences. The total score is reported and ranges from 0 (no consequences) to 50 (each of the possible consequences experienced).
  score on a scale | 14.7 (8.0) | 20.3 (7.3) | 16.0 (10.3) | 15.0 (8.7) | 16.8 (8.9)
Alcohol Use Disorder Identification Test (AUDIT) Score [Mean (Standard Deviation); unit: score on a scale] — The AUDIT is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. The scale ranges from 0 to 40; a score of 8 or more is considered to indicate hazardous or harmful alcohol use.
  score on a scale | 9.7 (3.8) | 13.9 (6.4) | 12.1 (6.5) | 12.9 (7.2) | 12.5 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: The average number of participants enrolled per week over the course of the study.
Time Frame: over the course of the study, approximately 8 months
Measure: Mean (Full Range); unit: average participants per week
Groups:
- Total Enrolled Patient Sample: All feasibility trial arms
Arm/Group | Total Enrolled Patient Sample
Number analyzed (Participants) | 75
average participants per week | 6.25 [3 to 9]

2. Primary Outcome: Drinker Inventory of Consequences (DrInC) Score
Description: The DrInC is a self-administered 50-item questionnaire designed to measure adverse consequences of alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. Scales are combined to assess total adverse consequences, with higher scores indicating more adverse consequences. This is a mean and standard deviation of the number of consequences suffered by participants since enrollment. The total DrInC score is reported where is 0 (no consequences) to 50 (every consequence experienced).
Time Frame: 6 weeks, 3 months, 6 months
Population: Participants who completed the specific follow up time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on the total scale
Groups:
- BNI Only: In the BNI arm, patients will receive a 5-30 minute brief negotiational intervention about their alcohol use as well as the standard discharge information and instructions.
  Brief Negotiational Intervention: This is a 5-10 minute conversation using the principles of motivational interviewing between the healthcare practioner and the patient to motivate the patient to identify at risk alcohol use and through self-empowerment create a plan to decrease alcohol use.
Arm/Group | Usual Care | BNI Only | BNI Plus Standard Booster | BNI Plus Personalized Booster
Number analyzed (Participants) | 10 | 21 | 24 | 20
score on the total scale
  6 weeks: number analyzed (Participants) | 9 | 15 | 17 | 19
  6 weeks | 0.2 (0.7) | 0.9 (1.8) | 1.9 (7.8) | 0.3 (0.9)
  3 months: number analyzed (Participants) | 10 | 15 | 20 | 17
  3 months | 0.2 (0.6) | 0.4 (1.1) | 2.4 (8.5) | 0.7 (1.2)
  6 months: number analyzed (Participants) | 10 | 15 | 19 | 17
  6 months | 1.3 (3.5) | 1.2 (3.2) | 1.0 (3.1) | 0.7 (1.5)

3. Secondary Outcome: Retention Rates
Description: Reported as the number of participants who complete each follow up visit.
Time Frame: 6 weeks, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Groups:
- All Trial Participants: Total participants in the feasibility trial.
Arm/Group | Usual Care | BNI Only | BNI Plus Standard Booster | BNI Plus Personalized Booster | All Trial Participants
Number analyzed (Participants) | 10 | 21 | 24 | 20 | 75
Participants
  6 weeks | 9 | 15 | 17 | 19 | 60
  3 months | 10 | 15 | 20 | 17 | 62
  6 months | 10 | 17 | 19 | 17 | 63

4. Secondary Outcome: Alcohol Use Disorder Identification Test (AUDIT) Score
Description: The AUDIT is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. The scale ranges from 0 to 40; a score of 8 or more is considered to indicate hazardous or harmful alcohol use. Presented as the AUDIT mean score over the month prior to visit.
Time Frame: 6 weeks, 3 months, 6 months
Population: Only those participants who were retained on follow up were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | BNI Only | BNI Plus Standard Booster | BNI Plus Personalized Booster
Number analyzed (Participants) | 10 | 21 | 24 | 20
score on a scale
  6 weeks: number analyzed (Participants) | 9 | 15 | 17 | 19
  6 weeks | 0.33 (1.0) | 1.5 (2.5) | 1.9 (5.3) | 1.2 (1.4)
  3 months: number analyzed (Participants) | 10 | 15 | 20 | 17
  3 months | 0.7 (0.9) | 1.9 (1.3) | 2.9 (5.0) | 2.7 (1.4)
  6 months: number analyzed (Participants) | 10 | 17 | 19 | 17
  6 months | 4.4 (5.3) | 4.0 (4.1) | 3.3 (2.3) | 4.9 (2.6)

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Arm/Group | Usual Care | BNI Only | BNI Plus Standard Booster | BNI Plus Personalized Booster
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/21 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/21 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/21 | 0/24 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02828267/Prot_SAP_000.pdf